CLINICAL TRIAL: NCT04315662
Title: Effects of a Power Training at Two Different Loads on Muscle Quality and Functional Capacity in Women Aged 65-75.
Brief Title: Power Training on Muscle Quality and Functional Capacity in Women Aged 65-75.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad del Valle, Colombia (Other)
Collaborators: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CI5302
Record Dates: First submitted 2020-03-09; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Muscle Weakness; Muscle Loss
Keywords: Muscle quality; Functional capacity; Power training
MeSH Terms: conditions — Muscle Weakness; Muscular Atrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle power training with velocity loss (VL) of 10% (Experimental): Subjects followed a muscle power training for 8 weeks (2 sessions per week on alternate days) using the leg extension exercise, with similar relative intensity (50% 1RM). Between weeks one and four two series will be performed per session. Then the number of series will increase to three per session. The inter-set recovery period will be always of 2-min. Velocity loss will be of 10% (VL10) in each set.
  Interventions: Other: Muscle power training with velocity loss (VL) of 10%
- Muscle power training with velocity loss (VL) of 30% (Active Comparator): Subjects followed a muscle power training for 8 weeks (2 sessions per week on alternate days) using the leg extension exercise, with similar relative intensity (50% 1RM). Between weeks one and four two series will be performed per session. Then the number of series will increase to three per session. The inter-set recovery period will be always of 2-min. Velocity loss will be of 30% (VL30) in each set.
  Interventions: Other: Muscle power training with velocity loss (VL) of 30%

INTERVENTIONS:
Other: Muscle power training with velocity loss (VL) of 10% — Subjects followed a muscle power training for 8 weeks (2 sessions per week on alternate days) using the leg extension exercise, with similar relative intensity (50% 1RM). Between weeks one and four two series will be performed per session. Then the number of series will increase to three per session. The inter-set recovery period will be always of 2-min. Velocity loss will be of 10% (VL10) in each set.
  Arms: Muscle power training with velocity loss (VL) of 10%
Other: Muscle power training with velocity loss (VL) of 30% — Subjects followed a muscle power training for 8 weeks (2 sessions per week on alternate days) using the leg extension exercise, with similar relative intensity (50% 1RM). Between weeks one and four two series will be performed per session. Then the number of series will increase to three per session. The inter-set recovery period will be always of 2-min. Velocity loss will be of 30% (VL30) in each set.
  Arms: Muscle power training with velocity loss (VL) of 30%

SUMMARY:
Muscle power training has proven to be an effective intervention to prevent sarcopenia and frailty in old people. In the last decade, new concepts related to the functionality of old people have been generated, such as muscle quality and functional capacity.

The power training consists of rapid movements of short duration that imply a more specialized neuromuscular response and that improve the functional response reflected in activities of daily life that demand a certain manifestation of muscular power (stand up of a chair, climbing stairs, rebalance, accelerate suddenly, among others). Therefore, it is important to investigate the dose-response relationships in power training in older people and establish how possible improvements in muscle quality can be reflected in functional capacity.

The aim of this study is to compare the effects of power training at two different loads on muscle quality and functional capacity in women aged 65-75

DETAILED DESCRIPTION:
Fifty-six women will be randomly assigned to one of two muscle power training supervised for a physical activity instructor with different velocity loss (VL) thresholds: 10% (VL10) and 30% (VL30). Subjects followed a muscle power training for 8 weeks (2 sessions per week on alternate days) using the leg extension exercise, with similar relative intensity (50% 1RM). Between weeks one and four two series will be performed per session. Then the number of series will increase to three per session. The inter-set recovery period will be always of 2-min.

Before and after the muscle power training the following tests will be performed: 1) measure of body composition with dual-energy x-ray absorptiometry for determining the lean mass of thighs; 2) three functional test (chair stand test, time up go test with cognitive task and gait speed test); 3)Progressive loading test in a leg extension machine until finding the mean muscle power corresponding to 50% of 1RM (speed of concentric phase of 6.67 ± 0.04 m/s measured using a camera-based optoelectronic system).

ELIGIBILITY:
Inclusion Criteria:

* Women 65 to 75 years.
* Healthy volunteers.
* Have not perform muscle power training in the last six months.

Exclusion Criteria:

* History of asthma.
* History of uncontrolled diabetes.
* History of uncontrolled hypertension.
* History of cardiovascular disease.
* History of coronary heart disease.
* Smoker.
* Arrhythmias.
* Personal history of surgical procedures in the last three months.
* Uncontrolled non-communicable diseases.
* Psychological, sensitive, cognitive, neuromotor and/or osteo-muscular conditions that may affect participation in an exercise program.
* Under medical treatment with anticoagulants, bronchodilators, and/or steroids.

Ages: 65 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-02-11 (Estimated)

PRIMARY OUTCOMES:
Change on muscle quality: obtained by measuring mean leg extension power divided by muscle mass of thighs | Baseline and after 8 weeks
  The muscle quality will be obtained by measuring mean leg extension power divided by muscle mass of thighs (measured by dual-energy x-ray absorptiometry)

SECONDARY OUTCOMES:
Change on chair stand test | Baseline and after 8 weeks
  Participants stand up straight as quickly as they can five times, without stopping in between. After standing up each time, subjects will sit down and then stand up again. They will keep their arms folded across their chest. The examiner will be timing with a stopwatch.
Change on time up go test with cognitive task | Baseline and after 8 weeks
  The participant stands up from a chair, walks to the mark 3 m away, turns around, returns to the chair, and sits down again. The participants walk safely, as fast as possible. While walking, the participant counts backward in threes from a randomly chosen start number between 60 and 100 to avoid a learning effect.
Change on gait speed test | Baseline and after 8 weeks
  Participants walk a 4-m marked course at their usual walking pace, with the examiner timing their walk with a stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Santiago A Arboleda, Ph.D., Principal Investigator — Universidad del Valle, Cali, Colombia.
Locations (1):
- Universidad del Valle, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No